CLINICAL TRIAL: NCT00618137
Title: Longitudinal Assessment of Clinical and Molecular Pathology of Chronic Obstructive Lung Disease and the Possible Influence of Inert Dusts in Working Volunteers of the Greater Vienna Area
Brief Title: Inert Dusts and Pathology of Chronic Obstructive Pulmonary Disease
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Rolf Ziesche, Associated Professor of Medicine, Medical University of Vienna
Other Study IDs: COPD-AUVA
Record Dates: First submitted 2008-02-05; First posted 2008-02-18 (Estimated); Last update posted 2012-08-24 (Estimated); Status verified 2012-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Chronic obstructive pulmonary disease; Gene expression profiling; Inert dusts; Natural course; Prospective assessment
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Transbronchial lung biopsies Blood serum
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The main objective of the study is the exploration of the natural course of COPD and its biological background. To this end, active workers without COPD and workers in functional classes GOLD 0-III are investigated by a combined clinical and molecular approach. The study has been designed as a prospective, intraindividual pilot in 160 male or female volunteers of the greater Vienna Area over a period of three years for each individual volunteer.

DETAILED DESCRIPTION:
Primary endpoint Combined assessment of clinical and molecular data obtained in three sequential study visits over an investigative period of 36 months for each individual; this includes, in particular, the identification of single and clustered gene functions connected to deterioration or stability of pulmonary function at the end of the observation period.

Secondary endpoints Assessment of occupational and environmental exposure to primarily inert fine dusts in a random subset of the strata by means of 24h-measurement of quantity and quality of fine dust inhalation; Influence of intensified exposure to fine dusts due to occupational conditions; Development of lung function in the five different study groups (see below), particularly changes from one GOLD class into the next class;

Definition of Study Groups:

Group 1 (Control):

Healthy volunteers, age 18 to 35 yr, never smokers (n=20).

Group 2 (preferentially taxi or bus drivers; COPD °0):

Working men/women, age 18 to 65 yr, preferentially taxi drivers or bus drivers or comparable occupational burden, current smokers or ex-smokers, with symptoms suggestive of COPD, yet regular lung function test at rest at the time of study entry, no signs of significant other diseases, in particular no signs of cardiovascular disease (n=35).

Group 3 (preferentially taxi or bus drivers; COPD °I-III):

Working men/women, preferentially taxi drivers or bus drivers or comparable occupational burden, age 35 to 65 yr, current smokers or ex-smokers, with symptoms of COPD, and abnormal lung function at rest at the time of study entry, no signs of significant other diseases, in particular no signs of cardiovascular disease (n=35).

Group 4 (Welder; COPD °0):

Working men/women, active welders or comparable occupational burden, age 35 to 65 yr, current smoker or ex-smoker, with symptoms suggestive of COPD, yet regular lung function test at rest, no signs of significant other diseases, in particular no signs of cardiovascular disease (n=35).

Group 5 (Welder; COPD °I-III):

Working men/women, active welders or comparable occupational burden, age 35 to 65 yr, current smoker or ex-smoker, with symptoms of COPD and abnormal lung function at rest at the time of study entry, no signs of significant other diseases, in particular no signs of cardiovascular disease (n=35).

Exclusion criteria:

* COPD °IV
* Bronchial asthma
* Major cardiovascular diseases, in particular stroke and myocardial infarction with reduced cardiac function
* Age > 65 years
* Acute or chronic bronchial infections, in particular bronchiectasis
* Cancer

Study investigations

Visit 1 Visit 2 Visit 3 Clinical investigation x x x Blood drawing for laboratory testing x x x Spirometry x x x Body plethysmography x x x Spiro-Ergometry x x x CT Thorax x x x Bronchoscopy with transbronchial biopsy x x x Gene profiling x x x

ELIGIBILITY:
Inclusion Criteria:

* COPD °0-III
* Workers of the greater Vienna Area
* Current smokers or ex-smokers

Exclusion Criteria:

* COPD °IV
* Bronchial asthma
* Major cardiovascular diseases, in particular stroke and myocardial infarction with reduced cardiac function
* Age > 65 years
* Acute or chronic bronchial infection, in particular bronchiectasis
* Cancer

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample of workers from the greater Vienna area
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2007-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lutz H Block, MD, Principal Investigator — Medical University of Vienna; Rolf Ziesche, MD, Study Director — Medical University of Vienna
Locations (1):
- Department of Pulmonary Medicine, Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Derived] Samaha E, Vierlinger K, Weinhappel W, Godnic-Cvar J, Nohammer C, Koczan D, Thiesen HJ, Yanai H, Fraifeld VE, Ziesche R. Expression Profiling Suggests Loss of Surface Integrity and Failure of Regenerative Repair as Major Driving Forces for Chronic Obstructive Pulmonary Disease Progression. Am J Respir Cell Mol Biol. 2021 Apr;64(4):441-452. doi: 10.1165/rcmb.2020-0270OC. PMID 33524306